CLINICAL TRIAL: NCT05485207
Title: T3STOPBPS: Open Label Clinical Trial of Transvaginal Trigone Treatment (T3) With Botulinum Toxin A (BTA) for Interstitial Cystitis / Bladder Pain Syndrome (IC/BPS)
Brief Title: Transvaginal Botulinum Toxin A for Interstitial Cystitis / Bladder Pain Syndrome
Acronym: T3STOPBPS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: McCormick and Gabilan Faculty Fellowship Award (Unknown)
Responsible Party: Principal Investigator, Amy Diane Dobberfuhl, Assistant Professor of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-58532
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: IC/BPS
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Transvaginal Botulinum Toxin A (BTA) injection (Experimental): Botulinum toxin A (Botox® 100 units) will be injected into the detrusor muscle of the bladder by inserting a needle through the anterior vaginal wall.
  Interventions: Drug: Transvaginal botulinum toxin A (BTA) injection

INTERVENTIONS:
Drug: Transvaginal botulinum toxin A (BTA) injection — Botulinum toxin A (Botox® 100 units) will be injected into the detrusor muscle of the bladder by inserting a needle through the anterior vaginal wall.
  Other Names: Botox® 100 units

SUMMARY:
Interstitial cystitis / bladder pain syndrome (IC/BPS) is a debilitating condition that affects millions of women in the United States. Women suffer from recurring pelvic pain, bladder pressure, painful bladder, urinary frequency (needing to go often) and urgency (feeling a strong need to go). Women are five times more likely to suffer from IC/BPS than men. IC/BPS is a common cause of painful bladder after excluding urinary tract infection. About one-third of women resort to opioids, thus contributing to the current opioid crisis. Sadly, there are no durable treatments and the majority of therapies are not FDA-approved for IC/BPS.

DETAILED DESCRIPTION:
Botulinum toxin A (BTA) injected into the bladder wall off-label for the IC/BPS indication has been effective in many women. Unfortunately most women cannot get BTA injection without general anesthesia due to pain from cystoscopy (small camera placed in the bladder). Dr. Dobberfuhl and her team created the transvaginal trigone treatment (T3) approach. Dr. Dobberfuhl was the first investigator in the world to complete a clinical trial of 31 injections of T3 BTA through the vaginal approach, for a non-painful condition, overactive bladder.

The T3STOPBPS study is an open label dose-escalation clinical study of BTA, for women with refractory IC/BPS. BTA is injected through the vaginal wall using a simple technique, the T3 approach, without the need for anesthesia or cystoscopy. The T3 BTA injection procedure has been well tolerated. The T3STOPBPS study will generate data needed for NIH R01 funding which will 1. Bring us closer to making T3 BTA available to women with IC/BPS, 2. Identify neuropeptide (pain) signaling targets for new IC/BPS therapies, and 3. Improve our understanding of fNIRS brain connectivity associated with IC/BPS treatment success.

Twelve patients will be recruited from the clinical practice of Dr. Dobberfuhl to undergo 50 unit T3 BTA injection at baseline. Psychometrically validated questionnaires (AUASS, ICIQ FLUTS, SF12, OLS ICSI / ICPI), voiding diaries, fNIRS and whole urine will be obtained at baseline (pre-treatment), 6 and 12 weeks after T3 BTA. Noninvasive fNIRS brain testing will be performed in collaboration with Dr. Hosseini, which will assess changes in cerebral connectivity from baseline. Whole urine will assess changes in neuropeptide molecular signaling using bulk RNA sequencing following T3 BTA treatment. RNA sequencing will be correlated with our single cell sequencing bladder biopsy data in IC/BPS. Following 50 unit T3 BTA injection, after the 12 week study visit, subjects will be offered dose escalation to 100 units if they do not achieve >50% improvement in PGIC. Milestone for T3 BTA efficacy will be met if >50% improvement is achieved in PGIC versus baseline. Subjects will be eligible for repeat BTA injection when they report less than 50% improvement in symptoms according to the patient global impression of change (PGIC) scale after the 12 week study visit. This will help us understand how long the effect of the BTA lasts, which is typically 3 to 12 months with the traditional cystoscopic route of delivery. A new consent form will be signed at the time of repeat injection.

ELIGIBILITY:
Inclusion Criteria:

* Females with IC/BPS
* Females who are considering intradetrusor BTA chemodenervation for the treatment of refractory IC/BPS

Exclusion Criteria:

* Involvement in other studies with potentially overlapping indications or symptoms
* Patients who are unable to undergo a transvaginal intervention as a result of anatomic barriers or discomfort will be excluded from enrollment
* patients known to be pregnant or breastfeeding
* Known allergy to BTA injection therapy or lidocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Patient Global Impression of Change (PGIC) scale | Baseline through week 12
  Patients will be classified as treatment success if they achieve our primary efficacy outcome of a >50% improvement in the Patient Global Impression of Change (PGIC) scale

SECONDARY OUTCOMES:
Change from baseline in American Urological Association Symptom Score (AUASS) | Baseline through week 12
  American Urological Association Symptom Score
Change from baseline in International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ FLUTS) | Baseline through week 12
  International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms
Change from baseline in Short Form 12-item Survey (SF12) | Baseline through week 12
  Short Form 12-item Survey
Change from baseline in O'Leary Sant (OLS) Symptom Score [Interstitial Cystitis Symptom Index (ICSI) / Interstitial Cystitis Problem Index (ICPI)] | Baseline through week 12
  O'Leary Sant Symptom Score (Interstitial Cystitis Symptom Index / Interstitial Cystitis Problem Index)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Dobberfuhl, M.D., Principal Investigator — Stanford University
Locations (1):
- Urology Clinic (Stanford University), 1000 Welch Road, Suite 100, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syan R, Briggs MA, Olivas JC, Srivastava S, Comiter CV, Dobberfuhl AD. Transvaginal ultrasound guided trigone and bladder injection: A cadaveric feasibility study for a novel route of intradetrusor chemodenervation. Investig Clin Urol. 2019 Jan;60(1):40-45. doi: 10.4111/icu.2019.60.1.40. Epub 2018 Dec 24. PMID 30637360
- [Background] Dobberfuhl AD, van Uem S, Versi E. Trigone as a diagnostic and therapeutic target for bladder-centric interstitial cystitis/bladder pain syndrome. Int Urogynecol J. 2021 Dec;32(12):3105-3111. doi: 10.1007/s00192-021-04878-9. Epub 2021 Jun 22. PMID 34156506
- [Background] Dobberfuhl AD. Pathophysiology, assessment, and treatment of overactive bladder symptoms in patients with interstitial cystitis/bladder pain syndrome. Neurourol Urodyn. 2022 Nov;41(8):1958-1966. doi: 10.1002/nau.24958. Epub 2022 May 24. PMID 35607890